CLINICAL TRIAL: NCT05103332
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Zilebesiran Used as Add-on Therapy in Patients With Hypertension Not Adequately Controlled by a Standard of Care Antihypertensive Medication
Brief Title: Zilebesiran as Add-on Therapy in Patients With Hypertension Not Adequately Controlled by a Standard of Care Antihypertensive Medication (KARDIA-2)
Acronym: KARDIA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-AGT01-003; 2021-003776-13 (EudraCT Number)
Record Dates: First submitted 2021-10-22; First posted 2021-11-02 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
Keywords: High blood pressure; Hypertension; Hypertensive; siRNA; Angiotensinogen; AGT
MeSH Terms: conditions — Hypertension | interventions — Indapamide; Amlodipine; olmesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Add-on to Indapamide) (Placebo Comparator): Following a 4-week run-in treatment on indapamide, 2.5 milligrams (mg), orally, once daily (QD), eligible participants were randomized to receive placebo matched to zilebesiran as a subcutaneous (SC) injection on Day 1 of 6-month double-blind (DB) treatment period as add-on therapy to indapamide. Participants received protocol-assigned background medication for 6 months, after which it was discontinued. Thereafter, participants will receive zilebesiran once every 6 months (Q6M) during the open-label extension (OLE) period. Upon implementation of Amendment 3, the OLE period was closed.
  Interventions: Drug: Indapamide; Drug: Placebo; Drug: Zilebesiran
- Zilebesiran (Add-on to Indapamide) (Experimental): Following a 4-week run-in treatment on indapamide, 2.5 mg, orally, QD, eligible participants were randomized to receive zilebesiran 600 mg, as a SC injection on Day 1 of 6-month DB treatment period as add-on therapy to indapamide. Participants received protocol-assigned background medication for 6 months, after which it was discontinued. Thereafter, participants will receive zilebesiran, Q6M during the OLE period. Upon implementation of Amendment 3, the OLE period was closed.
  Interventions: Drug: Indapamide; Drug: Zilebesiran
- Placebo (Add-on to Amlodipine) (Placebo Comparator): Following a 4-week run-in treatment on amlodipine, 5 mg, orally, QD, eligible participants were randomized to receive placebo matched to zilebesiran as a SC injection on Day 1 of 6-month DB treatment period as add-on therapy to amlodipine. Participants received protocol-assigned background medication for 6 months, after which it was discontinued. Thereafter, participants will receive zilebesiran Q6M during the OLE period. Upon implementation of Amendment 3, the OLE period was closed.
  Interventions: Drug: Amlodipine; Drug: Placebo; Drug: Zilebesiran
- Zilebesiran (Add-on to Amlodipine) (Experimental): Following a 4-week run-in treatment on amlodipine, 5 mg, orally, QD, eligible participants were randomized to receive zilebesiran 600 mg, as a SC injection on Day 1 of 6-month DB treatment period as add-on therapy to amlodipine. Participants received protocol-assigned background medication for 6 months, after which it was discontinued. Thereafter, participants will receive zilebesiran, Q6M during the OLE period. Upon implementation of Amendment 3, the OLE period was closed.
  Interventions: Drug: Amlodipine; Drug: Zilebesiran
- Placebo (Add-on to Olmesartan) (Placebo Comparator): Following a 4-week run-in treatment on olmesartan, 40 mg, orally, QD, (or 20 mg, orally, QD for participants with creatinine clearance ≤60 milliliters per minute [mL/min] at screening enrolled at sites outside of the United States [US] consistent with local labeling), eligible participants were randomized to receive placebo matched to zilebesiran as a SC injection on Day 1 of 6-month DB treatment period as add-on therapy to olmesartan. Participants received protocol-assigned background medication for 6 months, after which it was discontinued. Thereafter, participants will receive zilebesiran Q6M during the OLE period. Upon implementation of Amendment 3, the OLE period was closed.
  Interventions: Drug: Olmesartan; Drug: Placebo; Drug: Zilebesiran
- Zilebesiran (Add-on to Olmesartan) (Experimental): Following a 4-week run-in treatment on olmesartan, 40 mg, orally, QD, (or 20 mg, orally, QD for participants with creatinine clearance ≤60 mL/min at screening enrolled at sites outside of the US consistent with local labeling), eligible participants were randomized to receive zilebesiran 600 mg, as a SC injection on Day 1 of 6-month DB treatment period as add-on therapy to olmesartan. Participants received protocol-assigned background medication for 6 months, after which it was discontinued. Thereafter, participants will receive zilebesiran, Q6M during the OLE period. Upon implementation of Amendment 3, the OLE period was closed.
  Interventions: Drug: Olmesartan; Drug: Zilebesiran

INTERVENTIONS:
Drug: Indapamide — Indapamide administered orally
  Arms: Placebo (Add-on to Indapamide); Zilebesiran (Add-on to Indapamide)
Drug: Amlodipine — Amlodipine administered orally
  Arms: Placebo (Add-on to Amlodipine); Zilebesiran (Add-on to Amlodipine)
Drug: Olmesartan — Olmesartan administered orally
  Arms: Placebo (Add-on to Olmesartan); Zilebesiran (Add-on to Olmesartan)
Drug: Placebo — Placebo administered by SC injection
  Arms: Placebo (Add-on to Amlodipine); Placebo (Add-on to Indapamide); Placebo (Add-on to Olmesartan)
Drug: Zilebesiran — Zilebesiran administered by SC injection
  Other Names: ALN-AGT01

SUMMARY:
The purpose of this study is to evaluate the effect of zilebesiran on systolic and diastolic blood pressure and to characterize the pharmacodynamic (PD) effects and safety of zilebesiran as add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Office SBP at Screening as follows:

  1. ≥155 mmHg and ≤180 mmHg for patients with untreated hypertension
  2. ≥145 mmHg and ≤180 mmHg for patients on antihypertensive medications
* 24-hour mean SBP ≥130 mmHg and ≤160 mmHg by ABPM after at least 4 weeks of run-in

Exclusion Criteria:

* Secondary hypertension, orthostatic hypotension
* Elevated potassium <lower limit of normal (LLN) range or >5 milliequivalents per liter (mEq/L)
* Estimated glomerular filtration rate (eGFR) of <30 mL/min/1.73m^2
* Received an investigational agent within the last 30 days
* Type 1 diabetes mellitus, poorly controlled Type 2 diabetes mellitus, or laboratory evidence of diabetes during screening without known diagnosis of diabetes
* History of any cardiovascular event within 6 months prior to randomization
* History of intolerance to SC injection(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (101):
- United States (65):
  - Clinical Trial Site, Mesa, Arizona
  - Clinical Trial Site, Tempe, Arizona
  - Clinical Trial Site, Bell Gardens, California
  - Clinical Trials Site, Beverly Hills, California
  - Clinical Trial Site, Canoga Park, California
  - Clinical Trial Site, Carlsbad, California
  - Clinical Trial Site, Encinitas, California
  - Clinical Trial Site, Garden Grove, California
  - Clinical Trial Site, Hollywood, California
  - Clinical Trial Site, Huntington Beach, California
  - Clinical Trial Site, Irvine, California
  - Clinical Trial Site, Long Beach, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Mission Hills, California
  - Clinical Trial Site, Oceanside, California
  - Clinical Trial Site, Panorama City, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Santa Clarita, California
  - Clinical Trial Site, South Gate, California
  - Clinical Trial Site, Tustin, California
  - Clinical Trial Site, Upland, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Coconut Creek, Florida
  - Clinical Trial Site, Coral Gables, Florida
  - Clinical Trial Site, Hollywood, Florida
  - Clinical Trial Site, Inverness, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Naples, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Pembroke Pines, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Winter Haven, Florida
  - Clinical Trial Site, Winter Park, Florida
  - Clinical Trial Site, Acworth, Georgia
  - Clinical Trial Site, Canton, Georgia
  - Clinical Trial Site, Columbus, Georgia
  - Clinical Trial Site, Savannah, Georgia
  - Clinical Trial Site, Louisville, Kentucky
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Southgate, Michigan
  - Clinical Trial Site, Jackson, Mississippi
  - Clinical Trial Site, Hazelwood, Missouri
  - Clinical Trial Site, Jefferson City, Missouri
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Greensboro, North Carolina
  - Clinical Trial Site, Monroe, North Carolina
  - Clinical Trial site, Winston-Salem, North Carolina
  - Clinical Trial Site, Norman, Oklahoma
  - Clinical Trial Site, Little River, South Carolina
  - Clinical Trial Site, Memphis, Tennessee
  - Clinical Trial Site, Amarillo, Texas
  - Clinical Trial Site, Coppell, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Lake Jackson, Texas
  - Clinical Trial Site, Plano, Texas
  - Clinical Trial Site, Sherman, Texas
  - Clinical Trial Site, Splendora, Texas
  - Clinical Trial Site, Stephenville, Texas
  - Clinical Trial Site, Tomball, Texas
  - Clinical Trial Site, Waco, Texas
  - Clinical Trial Site, Burke, Virginia
  - Clinical Trial Site, Kenosha, Wisconsin
- Canada (12):
  - Clinical Trial Site, Brampton, Ontario
  - Clinical Trial Site, Concord, Ontario
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Winnipeg, Ontario
  - Clinical Trial Site, Chicoutimi, Quebec
  - Clinical Trial Site, Lévis, Quebec
  - Clinical Trial Site, Pointe-Claire, Quebec
  - Clinical Trial Site, Québec, Quebec
  - Clinical Trial Site, Sherbrooke, Quebec
  - Clinical Trial Site, Trois-Rivières, Quebec
  - Clinical Trial Site, Québec
- Clinical Trial Site, Tartu, Estonia
- Clinical Trial Site, Frankfurt, Germany
- Clinical Trial Site, Riga, Latvia
- Lithuania (2):
  - Clinical Trial Site, Kaunas
  - Clinical Trial Site, Vilnius
- Poland (6):
  - Clinical Trial Site, Częstochowa
  - Clinical Trial Site, Gdansk
  - Clinical Trial Site, Katowice
  - Clinical Trial Site, Staszów
  - Clinical Trial Site, Warsaw
  - Clinical Trial Site, Wroclaw
- United Kingdom (13):
  - Clinical Trial Site, Bellshill, Lanarkshire
  - Clinical Trial Site, Carshalton
  - Clinical Trial Site, Edinburgh
  - Clinical Trial Site, Fowey
  - Clinical Trial Site, Glasgow
  - Clinical Trial Site, Lancashire Preston
  - Clinical Trial Site, Liskeard
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester
  - Clinical Trial Site, Newquay
  - Clinical Trial Site, Plymouth
  - Clinical Trial Site, Sheffield
  - Clinical Trial Site, Torpoint

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the United States (US) and/or the European Union (EU).
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Desai AS, Karns AD, Badariene J, Aswad A, Neutel JM, Kazi F, Park W, Stiglitz D, Makarova N, Havasi A, Zappe DH, Saxena M; KARDIA-2 Study Group. Add-On Treatment With Zilebesiran for Inadequately Controlled Hypertension: The KARDIA-2 Randomized Clinical Trial. JAMA. 2025 Jul 1;334(1):46-55. doi: 10.1001/jama.2025.6681. PMID 40434761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 78 clinical sites in North America (66=United States [US] & 12=Canada) & 24 clinical sites in Europe (10=United Kingdom [UK]) enrolled participants in this study. 663 participants who met eligibility criteria after run-in with protocol-assigned background medication (indapamide, amlodipine, olmesartan) were randomized to zilebesiran or placebo in double-blind (DB) period, with the option to receive zilebesiran in open-label extension period (OLE). 1 month=28 days for this study.
Pre-assignment Details: Before Protocol Amendment 3 (PA3), participants completing DB period could join a separate zilebesiran OLE study. Those completing DB before OLE study availability entered OLE period in this study to receive zilebesiran until transition. Others ineligible for OLE study/discontinued drug in DB could enter safety follow-up(SFU). With PA3, OLE period was closed & plans for OLE study canceled. Ongoing DB participants entered SFU at completion; those in OLE stopped treatment & transitioned to SFU.
Groups:
- DB Period: Placebo (Add-on to Indapamide): Participants were randomized to receive placebo matched to zilebesiran, as a subcutaneous (SC) injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to indapamide. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Zilebesiran (Add-on to Indapamide): Participants were randomized to receive zilebesiran, 600 milligrams (mg), as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to indapamide. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Placebo (Add-on to Amlodipine): Participants were randomized to receive placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to amlodipine. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Zilebesiran (Add-on to Amlodipine): Participants were randomized to receive zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to amlodipine. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Placebo (Add-on to Olmesartan): Participants were randomized to receive placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Zilebesiran (Add-on to Olmesartan): Participants were randomized to receive zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort]: Prior to Amendment 3, participants who completed the DB period before a separate OLE study was available, entered the OLE period of this study and received treatment with zilebesiran 600 mg SC q6M. Protocol-specified background antihypertensive treatment with indapamide was discontinued at the start of OLE period.
- DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort]: Prior to Amendment 3, participants who completed the DB period before a separate OLE study was available, entered the OLE period of this study and continued treatment with zilebesiran 600 mg SC q6M. Protocol-specified background antihypertensive treatment with indapamide was discontinued at the start of OLE period.
- DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort]: Prior to Amendment 3, participants who completed the DB period before a separate OLE study was available, entered the OLE period of this study and received treatment with zilebesiran 600 mg SC q6M. Protocol-specified background antihypertensive treatment with amlodipine was discontinued at the start of OLE period.
- DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort]: Prior to Amendment 3, participants who completed the DB period before a separate OLE study was available, entered the OLE period of this study and continued treatment with zilebesiran 600 mg SC q6M. Protocol-specified background antihypertensive treatment with amlodipine was discontinued at the start of OLE period.
- DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort]: Prior to Amendment 3, participants who completed the DB period before a separate OLE study was available, entered the OLE period of this study and received treatment with zilebesiran 600 mg SC q6M. Protocol-specified background antihypertensive treatment with olmesartan was discontinued at the start of OLE period.
- DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort]: Prior to Amendment 3, participants who completed the DB period before a separate OLE study was available, entered the OLE period of this study and continued treatment with zilebesiran 600 mg SC q6M. Protocol-specified background antihypertensive treatment with olmesartan was discontinued at the start of OLE period.
- DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort]; DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort]; DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort]: Prior to Amendment 3, participants who did not enter OLE period or who discontinued treatment (placebo) during DB period entered SFU period.
  Upon implementation of Amendment 3, participants who completed the DB period entered the SFU period directly, and those already in OLE period did not receive any additional study drug in OLE and transitioned to the SFU period.
- DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort]; DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort]; DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort]: Prior to Amendment 3, participants who did not enter OLE period or who discontinued treatment (zilebesiran) during DB period entered SFU period.
  Upon implementation of Amendment 3, participants who completed the DB period entered the SFU period directly, and those already in OLE period did not receive any additional study drug in OLE and transitioned to the SFU period.
Period: DB Period (6 Months=168 Days)
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide) | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine) | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan) | DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort]
Started | 65 | 65 | 120 | 120 | 146 | 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Modified Full Analysis Set (mFAS) (mFAS included all randomized participants who received any amount of study drug. Analysis was grouped according to the randomized treatment arm.) | 64 | 63 | 120 | 118 | 146 | 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Modified Safety Analysis Set (mSAS) (mSAS included all participants who received any amount of the study drug. Participants were grouped according to the treatment actually received. 1 participant randomized to Placebo (Olmesartan) received zilebesiran, hence, was considered in the Zilebesiran (Olmesartan) arm for safety analysis.) | 64 | 63 | 120 | 118 | 145 | 148 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 63 | 59 | 114 | 115 | 143 | 139 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 6 | 6 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Stopped Participation in the Study | 2 | 3 | 5 | 3 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: OLE Period (24 Months=672 Days)
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide) | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine) | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan) | DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort]
Started | 0 | 0 | 0 | 0 | 0 | 0 | 26 (Participants who completed the 6-month DB period and met the eligibility criteria as per the study plan before implementation of protocol amendment 3 entered the OLE period.) | 30 (Participants who completed the 6-month DB period and met the eligibility criteria as per the study plan before implementation of protocol amendment 3 entered the OLE period.) | 48 (Participants who completed the 6-month DB period and met the eligibility criteria as per the study plan before implementation of protocol amendment 3 entered the OLE period.) | 44 (Participants who completed the 6-month DB period and met the eligibility criteria as per the study plan before implementation of protocol amendment 3 entered the OLE period.) | 66 (Participants who completed the 6-month DB period and met the eligibility criteria as per the study plan before implementation of protocol amendment 3 entered the OLE period.) | 60 (Participants who completed the 6-month DB period and met the eligibility criteria as per the study plan before implementation of protocol amendment 3 entered the OLE period.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 29 | 47 | 42 | 63 | 56 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: SFU Period (6 Months=168 Days)
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide) | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine) | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan) | DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Indapamide Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Amlodipine Cohort] | DB (Placebo) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort] | DB (Zilebesiran) to SFU or OLE (Zilebesiran) to SFU [Olmesartan Cohort]
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 (Upon implementation of Amendment 3, all participants who had completed the DB period entered the SFU period, and those in the OLE period did not receive any additional study drug in OLE and entered the SFU period.) | 59 (Upon implementation of Amendment 3, all participants who had completed the DB period entered the SFU period, and those in the OLE period did not receive any additional study drug in OLE and entered the SFU period.) | 114 (Upon implementation of Amendment 3, all participants who had completed the DB period entered the SFU period, and those in the OLE period did not receive any additional study drug in OLE and entered the SFU period.) | 115 (Upon implementation of Amendment 3, all participants who had completed the DB period entered the SFU period, and those in the OLE period did not receive any additional study drug in OLE and entered the SFU period.) | 143 (Upon implementation of Amendment 3, all participants who had completed the DB period entered the SFU period, and those in the OLE period did not receive any additional study drug in OLE and entered the SFU period.) | 139 (Upon implementation of Amendment 3, all participants who had completed the DB period entered the SFU period, and those in the OLE period did not receive any additional study drug in OLE and entered the SFU period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 57 | 55 | 106 | 104 | 133 | 126
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 8 | 11 | 10 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 3 | 4 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Stopped Participation in the Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 7 | 6 | 5
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The mFAS included all randomized participants who received any amount of study drug. Analysis was grouped according to the randomized treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide) | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine) | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan) | Total
Number analyzed (Participants) | 64 | 63 | 120 | 118 | 146 | 147 | 658
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.2) | 57.9 (10.7) | 58.4 (9.8) | 57.6 (10.2) | 57.7 (10.6) | 59.3 (10.4) | 58.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 50 | 53 | 64 | 60 | 282
  Male | 39 | 33 | 70 | 65 | 82 | 87 | 376
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 27 | 27 | 37 | 47 | 59 | 225
  Not Hispanic or Latino | 36 | 35 | 93 | 81 | 98 | 88 | 431
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 4 | 4 | 8 | 13 | 3 | 32
  Black or African American | 14 | 16 | 41 | 39 | 39 | 38 | 187
  White | 48 | 41 | 74 | 71 | 93 | 106 | 433
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Multiple | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Not Reported | 1 | 0 | 1 | 0 | 0 | 0 | 2
24-hour Mean Systolic Blood Pressure (SBP) Assessed by Ambulatory Blood Pressure Monitoring (ABPM) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — SBP assessed by ABPM at baseline is reported here. 24-hour ABPM device was programmed to take readings every 20 minutes during day(6 am-9:59 pm) & every 30 minutes during night(10 pm-5:59 am). ABPM was considered adequate if: number of successful daytime readings were ≥33; number of successful nighttime readings were≥11; no more than 3 hours are not represented(3 sections of 60 minutes with 0 valid readings). To summarize 24-hour ABPM, hourly adjusted mean was calculated. Hourly adjusted mean was average blood pressure(BP) for each hour of the day. 24-hour mean was average of the hourly means.
  millimeter of mercury (mmHg) | 143.2 (8.4) | 143.4 (8.5) | 142.6 (8.2) | 143.3 (7.8) | 144.2 (8.3) | 143.6 (8.2) | 143.4 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Indapamide: Change From Baseline at Month 3 in 24-hour Mean SBP Assessed by ABPM - Censored Data
Description: 24-hour ABPM device was programmed to take readings every 20 minutes during day (6 am- 9:59 pm) and every 30 minutes during night (10 pm-5:59 am). ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; 3. no more than 3 hours are not represented (i.e.,3 sections of 60 minutes where 0 valid readings were obtained). To summarize 24-hour ABPM, the hourly adjusted mean was calculated. Hourly adjusted mean was the average BP for each hour of the day. The 24-hour mean was the average of the hourly means. Least squares (LS) mean and standard error (SE) were calculated using a mixed model repeated measures (MMRM) approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for SBP assessed using ABPM, while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline and Month 3
Population: The mFAS included all randomized participants who received any amount of study drug. Analysis was grouped according to the randomized treatment arm. Overall number analyzed is the number of participants with data available for analysis at Month 3.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 56 | 53
mmHg | -3.7 (1.56) | -15.7 (1.60)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Indapamide) vs DB Period: Zilebesiran (Add-on to Indapamide); A hierarchical testing procedure was used to control type I error at α=0.05 within each cohort & handle primary & key secondary endpoints analyses. Testing was then performed sequentially in order the endpoints are reported. Hierarchical testing sequence continued only when previous endpoint was statistically significant at nominal p-value < 0.05. Data for SBP, assessed using ABPM, while participants were on & within 2 weeks after stopping any escape medication were censored for this endpoint; Test type: Superiority; p < 0.0001, MMRM — MMRM: Fixed factors: treatment, visit, treatment-by-visit interaction, race (black/all other races); Covariates: Baseline (BA) 24-hour mean SBP using ABPM & BA estimated glomerular filtration rate (eGFR). Unstructured covariance matrix was used; Difference in LS Mean = -12.1, 95% CI 2-sided [-16.5 to -7.6], Standard Error of Mean 2.24 — LS Mean Difference between zilebesiran (add on to indapamide) and placebo (add on to indapamide), 95% CI was calculated using MMRM model

2. Primary Outcome: Amlodipine: Change From Baseline at Month 3 in 24-hour Mean SBP Assessed by ABPM - Censored Data
Description: 24-hour ABPM device was programmed to take readings every 20 minutes during day (6 am- 9:59 pm) and every 30 minutes during night (10 pm-5:59 am). ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; 3. no more than 3 hours are not represented (i.e.,3 sections of 60 minutes where 0 valid readings were obtained). To summarize 24-hour ABPM, the hourly adjusted mean was calculated. Hourly adjusted mean was the average BP for each hour of the day. The 24-hour mean was the average of the hourly means. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for SBP assessed using ABPM, while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 100 | 99
mmHg | -0.7 (1.14) | -10.5 (1.15)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Amlodipine) vs DB Period: Zilebesiran (Add-on to Amlodipine); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — MMRM model included treatment, visit, treatment-by-visit interaction, race (black or all other races) as fixed factors, with baseline 24-hour mean SBP assessed by ABPM and baseline eGFR as covariates. Unstructured covariance matrix was used; Difference in LS Mean = -9.7, 95% CI 2-sided [-12.9 to -6.6], Standard Error of Mean 1.61 — LS Mean Difference between zilebesiran (add on to amlodipine) and placebo (add on to amlodipine), 95% CI was calculated using MMRM model

3. Primary Outcome: Olmesartan: Change From Baseline at Month 3 in 24-hour Mean SBP Assessed by ABPM - Censored Data
Description: 24-hour ABPM device was programmed to take readings every 20 minutes during day (6 am- 9:59 pm) and every 30 minutes during night (10 pm-5:59 am). ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; 3. no more than 3 hours are not represented (i.e.,3 sections of 60 minutes where 0 valid readings were obtained). To summarize 24-hour ABPM, the hourly adjusted mean was calculated. Hourly adjusted mean was the average BP for each hour of the day. The 24-hour mean was average of the hourly means. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for SBP assessed using ABPM, while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- DB Period: Placebo (Add-on to Olmesartan): Participants were randomized to receive placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocolspecified background antihypertensive medication per Investigator judgement.
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 114 | 115
mmHg | -3.2 (1.34) | -7.7 (1.33)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Olmesartan) vs DB Period: Zilebesiran (Add-on to Olmesartan); A hierarchical testing procedure was used to control type I error at α=0.05 within each cohort & handle primary & key secondary endpoints analyses. Testing was then performed sequentially in order the endpoints are reported. Hierarchical testing sequence continued only when previous endpoint was statistically significant at nominal p-value < 0.05. Data for SBP, assessed using ABPM, while subjects were on & within 2 weeks after stopping any escape medication were censored for this endpoint; Test type: Superiority; p = 0.0183, MMRM — MMRM: Fixed factors: treatment, visit, treatment-by-visit interaction, race (black/all other races); Covariates: Baseline (BA) 24-hour mean SBP using ABPM & BA eGFR. Unstructured covariance matrix was used; Difference in LS Mean = -4.5, 95% CI 2-sided [-8.2 to -0.8], Standard Error of Mean 1.89 — LS Mean Difference between zilebesiran (add on to olmesartan) and placebo (add on to olmesartan), 95% CI was calculated using MMRM model

4. Secondary Outcome: Indapamide: Change From Baseline at Month 3 in Office SBP - Censored Data
Description: The mean office BP in the sitting position was used for the analysis. Office BP in the sitting position was collected with a set of 4 replicates. The average of the last 3 replicates was calculated and used for analysis. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for office SBP assessed while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 55 | 58
mmHg | -0.8 (1.55) | -19.3 (1.52)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Indapamide) vs DB Period: Zilebesiran (Add-on to Indapamide); A hierarchical testing procedure was used to control type I error at α=0.05 within each cohort and handle primary and key secondary endpoints analyses. Testing was then performed sequentially in order the endpoints are reported. Hierarchical testing sequence continued only when previous endpoint was statistically significant at nominal p-value < 0.05. Data for office SBP assessed while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint; Test type: Superiority; p < 0.0001, MMRM — MMRM model included treatment, visit, treatment-by-visit interaction, race (black or all other races) as fixed factors, with baseline office SBP and baseline eGFR as covariates. Unstructured covariance matrix was used; Difference in LS Mean = -18.5, 95% CI 2-sided [-22.8 to -14.2], Standard Error of Mean 2.17 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Indapamide: Time-adjusted Change From Baseline Through Month 6 in 24-hour Mean SBP, Assessed by ABPM - All Collected Data
Description: Time-adjusted change was defined as the area under the curve (AUC) of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for SBP assessed by ABPM, were included in the analysis for this endpoint.
Time Frame: Baseline through Month 6
Population: The mFAS included all randomized participants who received any amount of study drug. Analysis was grouped according to the randomized treatment arm. Overall number analyzed is the number of participants with data available for analysis at Month 6.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 57 | 53
mmHg | -4.6 (1.30) | -15.6 (1.35)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Indapamide) vs DB Period: Zilebesiran (Add-on to Indapamide); A hierarchical testing procedure was used to control type I error at α=0.05 within each cohort and handle primary and key secondary endpoints analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at nominal p-value < 0.05. All collected data for SBP assessed by ABPM, were included in the analysis for this endpoint; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -11, 95% CI 2-sided [-14.7 to -7.3], Standard Error of Mean 1.88 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Indapamide: Time-adjusted Change From Baseline Through Month 6 in Office SBP - All Collected Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for office SBP were included in the analysis for this endpoint.
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 60 | 58
mmHg | -4.5 (1.16) | -18.1 (1.18)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Indapamide) vs DB Period: Zilebesiran (Add-on to Indapamide); A hierarchical testing procedure was used to control type I error at α=0.05 within each cohort and handle primary and key secondary endpoints analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at nominal p-value < 0.05. All collected data for office SBP were included in the analysis for this endpoint; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; Difference in LS Mean = -13.6, 95% CI 2-sided [-16.9 to -10.3], Standard Error of Mean 1.66 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Indapamide: Percentage of Participants With 24-hour Mean SBP <130 mmHg and/or Reduction From Baseline ≥20 mmHg Assessed by ABPM Without Escape Antihypertensive Medications at Month 6
Description: 24-hour ABPM device was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly adjusted mean was the average of BP for each hour of the day. The 24-hour mean was average of the hourly means.
Time Frame: Month 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 57 | 53
percentage of participants | 14.0 | 64.2
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Indapamide) vs DB Period: Zilebesiran (Add-on to Indapamide); A hierarchical testing procedure was used to control type I error at α=0.05 within each cohort and handle primary and key secondary endpoints analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at nominal p-value < 0.05; Test type: Superiority; p < 0.0001, Regression, Logistic — Logistic regression model included treatment and race (black or all other races) as factors and baseline 24-hour mean SBP and baseline eGFR as covariates; Odds Ratio (OR) = 12.39, 95% CI 2-sided [4.61 to 33.29]

8. Secondary Outcome: Indapamide: Change From Baseline at Month 3 in 24-hour Mean Diastolic Blood Pressure (DBP), Assessed by ABPM - Censored Data
Description: 24-hour ABPM device was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly adjusted mean was the average BP for each hour of the day. The 24-hour mean was average of the hourly means. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for DBP assessed using ABPM, while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 56 | 53
mmHg | -1.3 (0.87) | -9.1 (0.89)

9. Secondary Outcome: Indapamide: Change From Baseline at Month 3 in Office DBP - Censored Data
Description: The mean office BP in the sitting position was used for the analysis. Office BP in the sitting position was collected with a set of 4 replicates. The average of the last 3 replicates was calculated and used for analysis. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for office DBP assessed while participants were on and within 2 weeks after stopping any escape medication was censored for this endpoint.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 55 | 58
mmHg | -0.2 (1.03) | -10.5 (1.01)

10. Secondary Outcome: Indapamide: Time-adjusted Change From Baseline Through Month 3 in 24-hour Mean SBP and DBP, Assessed by ABPM - Censored Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for SBP and DBP, assessed using ABPM, while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 56 | 53
mmHg
  24-hour Mean SBP | -2.5 (1.22) | -15.4 (1.26)
  24-hour Mean DBP | -0.9 (0.76) | -8.7 (0.78)

11. Secondary Outcome: Indapamide: Time-adjusted Change From Baseline in Office SBP and DBP Through Month 3 - Censored Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for office SBP and DBP, while participants were on and within 2 weeks after stopping any escape medication were censored for this endpoint.
Time Frame: Baseline through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 55 | 58
mmHg
  Office SBP | -2.5 (1.35) | -17.2 (1.34)
  Office DBP | -0.7 (0.78) | -9.2 (0.77)

12. Secondary Outcome: Indapamide: Change From Baseline at Month 6 in 24-hour Mean SBP and DBP, Assessed by ABPM - All Collected Data
Description: 24-hour ABPM device was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly adjusted mean was the average BP for each hour of the day. The 24-hour mean was average of the hourly means. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for SBP and DBP assessed by ABPM are included in the analysis for this endpoint.
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 57 | 53
mmHg
  24-hour Mean SBP | -5.8 (1.68) | -16.1 (1.74)
  24-hour Mean DBP | -3.2 (1.07) | -8.0 (1.11)

13. Secondary Outcome: Indapamide: Change From Baseline at Month 6 in Office SBP and DBP - All Collected Data
Description: The mean office BP in the sitting position was used for the analysis. Office BP in the sitting position was collected with a set of 4 replicates. The average of the last 3 replicates was calculated and used for analysis. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for office SBP and DBP, were included in the analysis for this endpoint.
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 60 | 58
mmHg
  Office SBP | -7.2 (1.82) | -15.5 (1.84)
  Office DBP | -3.6 (1.13) | -7.8 (1.15)

14. Secondary Outcome: Indapamide: Time-adjusted Change From Baseline Through Month 6 in 24-hour Mean DBP, Assessed by ABPM - All Collected Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for DBP assessed by ABPM were included in the analysis for this endpoint.
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 57 | 53
mmHg | -2.3 (0.77) | -8.5 (0.80)

15. Secondary Outcome: Indapamide: Time-adjusted Change From Baseline Through Month 6 in Office DBP - All Collected Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for office DBP were included in the analysis for this endpoint.
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 60 | 58
mmHg | -2.0 (0.67) | -9.5 (0.67)

16. Secondary Outcome: Indapamide: Change From Baseline in Daytime and Nighttime SBP and DBP by ABPM at Each Visit - All Collected Data
Description: ABPM device was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33; 2. the number of successful nighttime readings were ≥11; and 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for daytime and nighttime SBP and DBP, assessed by ABPM, were included in the analysis for this endpoint.
Time Frame: Baseline, and Month 2, 3 and 6
Population: The mFAS included all randomized participants who received any amount of study drug. Analysis was grouped according to the randomized treatment arm. Number analyzed are unique number of participants out of all the assessed participants who were evaluable for the specified category. Different participants may have contributed data for each category.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 64 | 63
mmHg
  Change in Daytime Mean SBP at Month 2: number analyzed (Participants) | 61 | 54
  Change in Daytime Mean SBP at Month 2 | -1.8 (1.54) | -15.9 (1.63)
  Change in Daytime Mean SBP at Month 3: number analyzed (Participants) | 61 | 54
  Change in Daytime Mean SBP at Month 3 | -5.3 (1.59) | -15.9 (1.68)
  Change in Daytime Mean SBP at Month 6: number analyzed (Participants) | 57 | 53
  Change in Daytime Mean SBP at Month 6 | -6.5 (1.64) | -16.4 (1.69)
  Change in Nighttime Mean SBP at Month 2: number analyzed (Participants) | 61 | 54
  Change in Nighttime Mean SBP at Month 2 | -0.5 (1.44) | -13.5 (1.53)
  Change in Nighttime Mean SBP at Month 3: number analyzed (Participants) | 61 | 54
  Change in Nighttime Mean SBP at Month 3 | -2.9 (1.94) | -14.2 (2.05)
  Change in Nighttime Mean SBP at Month 6: number analyzed (Participants) | 57 | 53
  Change in Nighttime Mean SBP at Month 6 | -4.3 (2.07) | -15.2 (2.14)
  Change in Daytime Mean DBP at Month 2: number analyzed (Participants) | 61 | 54
  Change in Daytime Mean DBP at Month 2 | -0.6 (0.95) | -8.6 (1.01)
  Change in Daytime Mean DBP at Month 3: number analyzed (Participants) | 61 | 54
  Change in Daytime Mean DBP at Month 3 | -2.6 (0.91) | -8.7 (0.96)
  Change in Daytime Mean DBP at Month 6: number analyzed (Participants) | 57 | 53
  Change in Daytime Mean DBP at Month 6 | -3.7 (1.09) | -7.7 (1.13)
  Change in Nighttime Mean DBP at Month 2: number analyzed (Participants) | 61 | 54
  Change in Nighttime Mean DBP at Month 2 | -0.4 (1.03) | -8.1 (1.10)
  Change in Nighttime Mean DBP at Month 3: number analyzed (Participants) | 61 | 54
  Change in Nighttime Mean DBP at Month 3 | -0.9 (1.12) | -8.6 (1.18)
  Change in Nighttime Mean DBP at Month 6: number analyzed (Participants) | 57 | 53
  Change in Nighttime Mean DBP at Month 6 | -1.8 (1.24) | -8.7 (1.28)

17. Secondary Outcome: Indapamide: Percent Change From Baseline in Serum Angiotensinogen (AGT)
Time Frame: Baseline, Week 2 and Months 1, 2, 3, 4, 5 and 6
Population: Modified Pharmacodynamic (PD) Analysis Set included all participants who received at least 1 full dose of study drug. All by-treatment analyses based on the Modified PD Analysis Set were grouped according to the treatment actually received. Number analyzed are unique number of participants out of all the assessed participants who were evaluable for the specified category. Different participants may have contributed data for each category.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo (Add-on to Indapamide): Participants received placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to indapamide. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- Zilebesiran (Add-on to Indapamide): Participants received zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to indapamide. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
Arm/Group | Placebo (Add-on to Indapamide) | Zilebesiran (Add-on to Indapamide)
Number analyzed (Participants) | 64 | 63
percent change
  Percent Change from Baseline at Week 2: number analyzed (Participants) | 62 | 60
  Percent Change from Baseline at Week 2 | 6.37 (29.27) | -91.99 (17.89)
  Percent Change from Baseline at Month 1: number analyzed (Participants) | 61 | 61
  Percent Change from Baseline at Month 1 | 1.90 (26.11) | -92.48 (28.49)
  Percent Change from Baseline at Month 2: number analyzed (Participants) | 61 | 60
  Percent Change from Baseline at Month 2 | 4.34 (32.24) | -95.50 (15.91)
  Percent Change from Baseline at Month 3: number analyzed (Participants) | 61 | 60
  Percent Change from Baseline at Month 3 | 4.86 (28.19) | -94.80 (17.89)
  Percent Change from Baseline at Month 4: number analyzed (Participants) | 61 | 59
  Percent Change from Baseline at Month 4 | 1.81 (30.86) | -92.28 (21.64)
  Percent Change from Baseline at Month 5: number analyzed (Participants) | 60 | 58
  Percent Change from Baseline at Month 5 | 1.23 (26.19) | -93.08 (17.07)
  Percent Change from Baseline at Month 6: number analyzed (Participants) | 59 | 56
  Percent Change from Baseline at Month 6 | 4.81 (26.12) | -91.92 (16.23)

18. Secondary Outcome: Amlodipine: Change From Baseline at Month 3 in Office SBP - Censored Data
Description: as for outcome 4
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 103 | 112
mmHg | -1.4 (1.20) | -11.5 (1.16)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Amlodipine) vs DB Period: Zilebesiran (Add-on to Amlodipine); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; Difference in LS Mean = -10.2, 95% CI 2-sided [-13.4 to -6.9], Standard Error of Mean 1.67 — [estimate comment as in outcome 2, analysis 1]

19. Secondary Outcome: Amlodipine: Time-adjusted Change From Baseline Through Month 6 in 24-hour Mean SBP, Assessed by ABPM - All Collected Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Treatment policy strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., all collected data for SBP assessed by ABPM, were included in the analysis for this endpoint.
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 102 | 103
mmHg | -1.8 (0.95) | -9.7 (0.97)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Amlodipine) vs DB Period: Zilebesiran (Add-on to Amlodipine); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -7.9, 95% CI 2-sided [-10.6 to -5.3], Standard Error of Mean 1.36 — [estimate comment as in outcome 2, analysis 1]

20. Secondary Outcome: Amlodipine: Time-adjusted Change From Baseline Through Month 6 in Office SBP - All Collected Data
Description: as for outcome 6
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 113 | 111
mmHg | -2.9 (0.82) | -11.5 (0.82)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Amlodipine) vs DB Period: Zilebesiran (Add-on to Amlodipine); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; Difference in LS Mean = -8.6, 95% CI 2-sided [-10.9 to -6.3], Standard Error of Mean 1.16 — [estimate comment as in outcome 2, analysis 1]

21. Secondary Outcome: Amlodipine: Percentage of Participants With 24-hour Mean SBP <130 mmHg and/or Reduction From Baseline ≥20 mmHg Assessed by ABPM Without Escape Antihypertensive Medications at Month 6
Description: as for outcome 7
Time Frame: Month 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 102 | 103
percentage of participants | 13.7 | 39.8
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Amlodipine) vs DB Period: Zilebesiran (Add-on to Amlodipine); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 5.08, 95% CI 2-sided [2.43 to 10.61]

22. Secondary Outcome: Amlodipine: Change From Baseline at Month 3 in 24-hour Mean DBP, Assessed by ABPM - Censored Data
Description: as for outcome 8
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 100 | 99
mmHg | -0.8 (0.63) | -6.6 (0.64)

23. Secondary Outcome: Amlodipine: Change From Baseline at Month 3 in Office DBP - Censored Data
Description: as for outcome 9
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 103 | 112
mmHg | -1.2 (0.84) | -6.2 (0.81)

24. Secondary Outcome: Amlodipine: Time-adjusted Change From Baseline Through Month 3 in 24-hour Mean SBP and DBP, Assessed by ABPM - Censored Data
Description: as for outcome 10
Time Frame: Baseline through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 100 | 99
mmHg
  24-hour Mean SBP | -0.9 (0.99) | -9.9 (1.00)
  24-hour Mean DBP | -0.7 (0.56) | -6.4 (0.57)

25. Secondary Outcome: Amlodipine: Time-adjusted Change From Baseline in Office SBP and DBP Through Month 3 - Censored Data
Description: as for outcome 11
Time Frame: Baseline through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 103 | 112
mmHg
  Office SBP | -1.4 (0.95) | -11.3 (0.96)
  Office DBP | -0.6 (0.60) | -6.1 (0.61)

26. Secondary Outcome: Amlodipine: Change From Baseline at Month 6 in 24-hour Mean SBP and DBP, Assessed by ABPM - All Collected Data
Description: as for outcome 12
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 102 | 103
mmHg
  24-hour Mean SBP | -3.0 (1.26) | -9.0 (1.26)
  24-hour Mean DBP | -1.6 (0.68) | -5.7 (0.68)

27. Secondary Outcome: Amlodipine: Change From Baseline at Month 6 in Office SBP and DBP - All Collected Data
Description: as for outcome 13
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 113 | 111
mmHg
  Office SBP | -5.8 (1.12) | -12.6 (1.13)
  Office DBP | -3.5 (0.74) | -6.7 (0.75)

28. Secondary Outcome: Amlodipine: Time-adjusted Change From Baseline Through Month 6 in 24-hour Mean DBP, Assessed by ABPM - All Collected Data
Description: as for outcome 14
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 102 | 103
mmHg | -1.1 (0.53) | -6.2 (0.54)

29. Secondary Outcome: Amlodipine: Time-adjusted Change From Baseline Through Month 6 in Office DBP - All Collected Data
Description: as for outcome 15
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 113 | 111
mmHg | -1.4 (0.52) | -6.2 (0.53)

30. Secondary Outcome: Amlodipine: Change From Baseline in Daytime and Nighttime SBP and DBP by ABPM at Each Visit - All Collected Data
Description: as for outcome 16
Time Frame: Baseline, and Month 2, 3 and 6
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 120 | 118
mmHg
  Change in Daytime Mean SBP at Month 2: number analyzed (Participants) | 112 | 108
  Change in Daytime Mean SBP at Month 2 | -2.2 (1.24) | -9.3 (1.26)
  Change in Daytime Mean SBP at Month 3: number analyzed (Participants) | 110 | 101
  Change in Daytime Mean SBP at Month 3 | -1.3 (1.14) | -11.0 (1.18)
  Change in Daytime Mean SBP at Month 6: number analyzed (Participants) | 102 | 103
  Change in Daytime Mean SBP at Month 6 | -3.3 (1.31) | -9.1 (1.31)
  Change in Nighttime Mean SBP at Month 2: number analyzed (Participants) | 112 | 108
  Change in Nighttime Mean SBP at Month 2 | 0.1 (1.31) | -7.3 (1.34)
  Change in Nighttime Mean SBP at Month 3: number analyzed (Participants) | 110 | 101
  Change in Nighttime Mean SBP at Month 3 | 0.1 (1.34) | -8.9 (1.39)
  Change in Nighttime Mean SBP at Month 6: number analyzed (Participants) | 102 | 103
  Change in Nighttime Mean SBP at Month 6 | -2.6 (1.48) | -8.8 (1.48)
  Change in Daytime Mean DBP at Month 2: number analyzed (Participants) | 112 | 108
  Change in Daytime Mean DBP at Month 2 | -0.8 (0.70) | -6.4 (0.72)
  Change in Daytime Mean DBP at Month 3: number analyzed (Participants) | 110 | 101
  Change in Daytime Mean DBP at Month 3 | -0.8 (0.66) | -7.2 (0.69)
  Change in Daytime Mean DBP at Month 6: number analyzed (Participants) | 102 | 103
  Change in Daytime Mean DBP at Month 6 | -1.5 (0.74) | -5.8 (0.74)
  Change in Nighttime Mean DBP at Month 2: number analyzed (Participants) | 112 | 108
  Change in Nighttime Mean DBP at Month 2 | -0.4 (0.76) | -5.2 (0.77)
  Change in Nighttime Mean DBP at Month 3: number analyzed (Participants) | 110 | 101
  Change in Nighttime Mean DBP at Month 3 | -0.4 (0.76) | -5.6 (0.79)
  Change in Nighttime Mean DBP at Month 6: number analyzed (Participants) | 102 | 103
  Change in Nighttime Mean DBP at Month 6 | -1.4 (0.84) | -5.8 (0.84)

31. Secondary Outcome: Amlodipine: Percent Change From Baseline in Serum AGT
Time Frame: Baseline, Week 2 and Months 1, 2, 3, 4, 5 and 6
Population: Modified PD Analysis Set included all participants who received at least 1 full dose of study drug. All by-treatment analyses based on the Modified PD Analysis Set were grouped according to the treatment actually received. Number analyzed are unique number of participants out of all the assessed participants who were evaluable for the specified category. Different participants may have contributed data for each category.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo (Add-on to Amlodipine): Participants received placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to amlodipine. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- Zilebesiran (Add-on to Amlodipine): Participants received zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to amlodipine. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
Arm/Group | Placebo (Add-on to Amlodipine) | Zilebesiran (Add-on to Amlodipine)
Number analyzed (Participants) | 120 | 118
percent change
  Percent Change from Baseline at Week 2: number analyzed (Participants) | 116 | 113
  Percent Change from Baseline at Week 2 | 2.67 (22.81) | -92.80 (15.99)
  Percent Change from Baseline at Month 1: number analyzed (Participants) | 117 | 112
  Percent Change from Baseline at Month 1 | 9.62 (35.83) | -95.35 (21.36)
  Percent Change from Baseline at Month 2: number analyzed (Participants) | 115 | 111
  Percent Change from Baseline at Month 2 | 11.23 (35.17) | -97.45 (8.59)
  Percent Change from Baseline at Month 3: number analyzed (Participants) | 113 | 109
  Percent Change from Baseline at Month 3 | 12.78 (34.90) | -96.37 (11.24)
  Percent Change from Baseline at Month 4: number analyzed (Participants) | 112 | 112
  Percent Change from Baseline at Month 4 | 12.42 (41.83) | -96.52 (8.41)
  Percent Change from Baseline at Month 5: number analyzed (Participants) | 111 | 107
  Percent Change from Baseline at Month 5 | 10.81 (37.94) | -93.87 (19.20)
  Percent Change from Baseline at Month 6: number analyzed (Participants) | 112 | 109
  Percent Change from Baseline at Month 6 | 9.51 (48.05) | -94.52 (9.37)

32. Secondary Outcome: Olmesartan: Change From Baseline at Month 3 in Office SBP - Censored Data
Description: as for outcome 4
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 117 | 121
mmHg | -2.6 (1.25) | -9.3 (1.23)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Olmesartan) vs DB Period: Zilebesiran (Add-on to Olmesartan); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 4, analysis 1]; Difference in LS Mean = -6.7, 95% CI 2-sided [-10.2 to -3.3], Standard Error of Mean 1.76 — [estimate comment as in outcome 3, analysis 1]

33. Secondary Outcome: Olmesartan: Time-adjusted Change From Baseline Through Month 6 in 24-hour Mean SBP, Assessed by ABPM - All Collected Data
Description: as for outcome 19
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 128 | 116
mmHg | -5.8 (0.99) | -7.6 (1.01)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Olmesartan) vs DB Period: Zilebesiran (Add-on to Olmesartan); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.2103, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -1.8, 95% CI 2-sided [-4.6 to 1.0], Standard Error of Mean 1.42 — [estimate comment as in outcome 3, analysis 1]

34. Secondary Outcome: Olmesartan: Time-adjusted Change From Baseline Through Month 6 in Office SBP - All Collected Data
Description: as for outcome 6
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 137 | 134
mmHg | -6.3 (0.81) | -10.8 (0.81)
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Olmesartan) vs DB Period: Zilebesiran (Add-on to Olmesartan); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; Difference in LS Mean = -4.5, 95% CI 2-sided [-6.8 to -2.3], Standard Error of Mean 1.14 — [estimate comment as in outcome 3, analysis 1]

35. Secondary Outcome: Olmesartan: Percentage of Participants With 24-hour Mean SBP <130 mmHg and/or Reduction From Baseline ≥20 mmHg Assessed by ABPM Without Escape Antihypertensive Medications at Month 6
Description: as for outcome 7
Time Frame: Month 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 128 | 116
percentage of participants | 17.2 | 25.9
Statistical Analysis 1: Comparison: DB Period: Placebo (Add-on to Olmesartan) vs DB Period: Zilebesiran (Add-on to Olmesartan); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.1230, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.87 to 3.23]

36. Secondary Outcome: Olmesartan: Change From Baseline at Month 3 in 24-hour Mean DBP, Assessed by ABPM - Censored Data
Description: as for outcome 8
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 114 | 115
mmHg | -1.4 (0.78) | -3.4 (0.78)

37. Secondary Outcome: Olmesartan: Change From Baseline at Month 3 in Office DBP - Censored Data
Description: as for outcome 9
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 117 | 121
mmHg | -2.0 (0.86) | -5.3 (0.85)

38. Secondary Outcome: Olmesartan: Time-adjusted Change From Baseline Through Month 3 in 24-hour Mean SBP and DBP, Assessed by ABPM - Censored Data
Description: as for outcome 10
Time Frame: Baseline through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 114 | 115
mmHg
  24-hour Mean SBP | -2.2 (1.12) | -5.3 (1.13)
  24-hour Mean DBP | -1.1 (0.63) | -2.3 (0.64)

39. Secondary Outcome: Olmesartan: Time-adjusted Change From Baseline in Office SBP and DBP Through Month 3 - Censored Data
Description: Time-adjusted change was defined as the AUC of BP change from baseline divided by the duration of the time period. LS mean and SE were calculated using a MMRM approach. Hypothetical strategy was used for the intercurrent event of using antihypertensive escape medication, i.e., data for office SBP and DBP, while participants were on and within 2 weeks after stopping any escape medication was censored for this endpoint.
Time Frame: Baseline through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 117 | 121
mmHg
  Office SBP | -2.4 (0.99) | -7.9 (0.97)
  Office DBP | -1.2 (0.65) | -3.8 (0.64)

40. Secondary Outcome: Olmesartan: Change From Baseline at Month 6 in 24-hour Mean SBP and DBP, Assessed by ABPM - All Collected Data
Description: as for outcome 12
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 128 | 116
mmHg
  24-hour Mean SBP | -9.2 (1.24) | -8.3 (1.29)
  24-hour Mean DBP | -5.2 (0.73) | -4.3 (0.76)

41. Secondary Outcome: Olmesartan: Change From Baseline at Month 6 in Office SBP and DBP - All Collected Data
Description: as for outcome 13
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 137 | 134
mmHg
  Office SBP | -11.9 (1.33) | -12.4 (1.34)
  Office DBP | -7.0 (0.76) | -7.1 (0.76)

42. Secondary Outcome: Olmesartan: Time-adjusted Change From Baseline Through Month 6 in 24-hour Mean DBP, Assessed by ABPM - All Collected Data
Description: as for outcome 14
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 128 | 116
mmHg | -3.1 (0.58) | -3.5 (0.59)

43. Secondary Outcome: Olmesartan: Time-adjusted Change From Baseline Through Month 6 in Office DBP - All Collected Data
Description: as for outcome 15
Time Frame: Baseline through Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 137 | 134
mmHg | -3.5 (0.53) | -5.8 (0.52)

44. Secondary Outcome: Olmesartan: Change From Baseline in Daytime and Nighttime SBP and DBP by ABPM at Each Visit - All Collected Data
Description: as for outcome 16
Time Frame: Baseline, and Month 2, 3 and 6
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 146 | 147
mmHg
  Change in Daytime Mean SBP at Month 2: number analyzed (Participants) | 132 | 128
  Change in Daytime Mean SBP at Month 2 | -1.0 (1.39) | -3.3 (1.41)
  Change in Daytime Mean SBP at Month 3: number analyzed (Participants) | 133 | 129
  Change in Daytime Mean SBP at Month 3 | -3.7 (1.29) | -8.5 (1.31)
  Change in Daytime Mean SBP at Month 6: number analyzed (Participants) | 128 | 116
  Change in Daytime Mean SBP at Month 6 | -8.8 (1.29) | -8.3 (1.34)
  Change in Nighttime Mean SBP at Month 2: number analyzed (Participants) | 132 | 128
  Change in Nighttime Mean SBP at Month 2 | -2.4 (1.53) | -2.7 (1.56)
  Change in Nighttime Mean SBP at Month 3: number analyzed (Participants) | 133 | 129
  Change in Nighttime Mean SBP at Month 3 | -5.3 (1.35) | -7.4 (1.37)
  Change in Nighttime Mean SBP at Month 6: number analyzed (Participants) | 128 | 116
  Change in Nighttime Mean SBP at Month 6 | -9.7 (1.35) | -8.4 (1.41)
  Change in Daytime Mean DBP at Month 2: number analyzed (Participants) | 132 | 128
  Change in Daytime Mean DBP at Month 2 | -0.5 (0.76) | -1.2 (0.77)
  Change in Daytime Mean DBP at Month 3: number analyzed (Participants) | 133 | 129
  Change in Daytime Mean DBP at Month 3 | -1.7 (0.76) | -3.9 (0.78)
  Change in Daytime Mean DBP at Month 6: number analyzed (Participants) | 128 | 116
  Change in Daytime Mean DBP at Month 6 | -5.0 (0.76) | -4.3 (0.79)
  Change in Nighttime Mean DBP at Month 2: number analyzed (Participants) | 132 | 128
  Change in Nighttime Mean DBP at Month 2 | -1.3 (0.86) | -1.4 (0.87)
  Change in Nighttime Mean DBP at Month 3: number analyzed (Participants) | 133 | 129
  Change in Nighttime Mean DBP at Month 3 | -2.6 (0.86) | -3.2 (0.87)
  Change in Nighttime Mean DBP at Month 6: number analyzed (Participants) | 128 | 116
  Change in Nighttime Mean DBP at Month 6 | -5.5 (0.85) | -4.2 (0.88)

45. Secondary Outcome: Olmesartan: Percent Change From Baseline in Serum AGT
Time Frame: Baseline, Week 2 and Months 1, 2, 3, 4, 5 and 6
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo (Add-on to Olmesartan): Participants received placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- Zilebesiran (Add-on to Olmesartan): Participants received zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
Arm/Group | Placebo (Add-on to Olmesartan) | Zilebesiran (Add-on to Olmesartan)
Number analyzed (Participants) | 144 | 148
percent change
  Percent Change from Baseline at Week 2: number analyzed (Participants) | 139 | 139
  Percent Change from Baseline at Week 2 | 8.08 (86.70) | -87.83 (35.99)
  Percent Change from Baseline at Month 1: number analyzed (Participants) | 143 | 140
  Percent Change from Baseline at Month 1 | 4.64 (28.05) | -92.61 (25.21)
  Percent Change from Baseline at Month 2: number analyzed (Participants) | 136 | 137
  Percent Change from Baseline at Month 2 | 4.87 (29.58) | -92.58 (29.50)
  Percent Change from Baseline at Month 3: number analyzed (Participants) | 137 | 136
  Percent Change from Baseline at Month 3 | 6.45 (28.36) | -92.98 (23.98)
  Percent Change from Baseline at Month 4: number analyzed (Participants) | 138 | 135
  Percent Change from Baseline at Month 4 | 4.62 (27.62) | -91.66 (25.44)
  Percent Change from Baseline at Month 5: number analyzed (Participants) | 139 | 131
  Percent Change from Baseline at Month 5 | 5.82 (31.65) | -91.14 (24.14)
  Percent Change from Baseline at Month 6: number analyzed (Participants) | 138 | 133
  Percent Change from Baseline at Month 6 | 1.93 (26.66) | -88.22 (41.42)

ADVERSE EVENTS:
Time Frame: Run-in: 4 weeks; DB Period (DBP): Day1 to Month6 (168 days); Zilebesiran (zil) Treatment Period: First zil dose to 6 months after last dose [Placebo (pbo)/Zil: Months 6 to 30 (672 days); Zil/Zil: Day1 to Month30 (840 days)]; SFU: 6 months (168 days); 1 month=28 days. Run-in: Participants eligible after run-in who received at least 1 dose of study drug in DBP, grouped per their background medication. DBP: mSAS; SFU: Participants from mSAS, grouped per last treatment in DB/OLE before SFU entry.
Description: As pre-specified in SAP, after DBP, AEs were reported by treatment sequence (Zil/Zil or pbo/Zil) for zilebesiran treatment period using All Zilebesiran Treated Set (Arms 10-15). Zil/Zil arm received zilebesiran in both DB & OLE. Hence, AEs' data for DB+OLE have been reported together. This set gives AEs for all participants receiving zilebesiran, including participants on zilebesiran during DB & continuing it after Month 6 & those on placebo in DB later & switching to zilebesiran after Month 6.
Groups:
- Run-in: Indapamide: Participants who cleared screening received open-label therapy with indapamide 2.5 mg orally once daily (QD) as their protocol-specified background antihypertensive medication during a Run-in period of at least 4 weeks.
- Run-in: Amlodipine: Participants who cleared screening received open-label therapy with amlodipine 5 mg orally QD as their protocol-specified background antihypertensive medication during a Run-in period of at least 4 weeks.
- Run-in: Olmesartan: Participants who cleared screening received open-label therapy with olmesartan 40 mg orally QD [or 20 mg orally QD for participants with creatinine clearance ≤ 60 mL/min at screening enrolled at sites outside of the US] as their protocol-specified background antihypertensive medication during a Run-in period of at least 4 weeks.
- DB Period: Placebo (Add-on to Indapamide): Participants received placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to indapamide. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Zilebesiran (Add-on to Indapamide): Participants received zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to indapamide. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Placebo (Add-on to Amlodipine): Participants received placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to amlodipine. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Zilebesiran (Add-on to Amlodipine): Participants received zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to amlodipine. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Placebo (Add-on to Olmesartan): Participants received placebo matched to zilebesiran, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB Period: Zilebesiran (Add-on to Olmesartan): Participants received zilebesiran, 600 mg, as a SC injection, on Day 1 of the 6-month DB treatment period as an add-on therapy to olmesartan. Starting at Month 3, additional conventional oral antihypertensives ("escape antihypertensive medications") may be added to the participant's protocol-specified background antihypertensive medication per Investigator judgement.
- DB (Placebo) to SFU [Indapamide Cohort]; DB (Placebo) to SFU [Amlodipine Cohort]; DB (Placebo) to SFU [Olmesartan Cohort]: Participants treated with placebo during DB period who did not enter the OLE period (prior to Amendment 3) or who discontinued treatment during the DB period entered the SFU period for safety monitoring.
  No treatment was administered in SFU.
- DB (Zilebesiran) to SFU or OLE to SFU [Indapamide Cohort]; DB (Zilebesiran) to SFU or OLE to SFU [Amlodipine Cohort]; DB (Zilebesiran) to SFU or OLE to SFU [Olmesartan Cohort]: Prior to Amendment 3, participants treated with zilebesiran who did not enter the OLE Period or who discontinued treatment (zilebesiran) during the DB period entered the SFU period for safety monitoring.
  Upon implementation of Amendment 3, participants who completed the DB period entered the SFU period directly. Participants who were already in OLE period (after completing treatment with zilebesiran/placebo in DB period) did not receive any additional study drug in OLE and transitioned to the SFU period for safety monitoring.
  No treatment was administered in SFU.
Arm/Group | Run-in: Indapamide | Run-in: Amlodipine | Run-in: Olmesartan | DB Period: Placebo (Add-on to Indapamide) | DB Period: Zilebesiran (Add-on to Indapamide) | DB Period: Placebo (Add-on to Amlodipine) | DB Period: Zilebesiran (Add-on to Amlodipine) | DB Period: Placebo (Add-on to Olmesartan) | DB Period: Zilebesiran (Add-on to Olmesartan) | DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort] | DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort] | DB (Placebo) to SFU [Indapamide Cohort] | DB (Zilebesiran) to SFU or OLE to SFU [Indapamide Cohort] | DB (Placebo) to SFU [Amlodipine Cohort] | DB (Zilebesiran) to SFU or OLE to SFU [Amlodipine Cohort] | DB (Placebo) to SFU [Olmesartan Cohort] | DB (Zilebesiran) to SFU or OLE to SFU [Olmesartan Cohort]
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/238 | 0/293 | 0/64 | 0/63 | 0/120 | 0/118 | 0/145 | 0/148 | 0/26 | 0/63 | 0/48 | 0/118 | 0/66 | 0/148 | 0/38 | 0/89 | 1/72 | 0/166 | 0/79 | 1/214
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/238 | 1/293 | 2/64 | 0/63 | 1/120 | 3/118 | 4/145 | 4/148 | 1/26 | 1/63 | 1/48 | 3/118 | 3/66 | 7/148 | 0/38 | 1/89 | 0/72 | 0/166 | 0/79 | 1/214
Other Adverse Events (participants affected / at risk) | 0/127 | 0/238 | 0/293 | 11/64 | 14/63 | 21/120 | 26/118 | 29/145 | 41/148 | 1/26 | 19/63 | 6/48 | 36/118 | 23/66 | 51/148 | 0/38 | 0/89 | 0/72 | 0/166 | 0/79 | 0/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in: Indapamide (N=127) | Run-in: Amlodipine (N=238) | Run-in: Olmesartan (N=293) | DB Period: Placebo (Add-on to Indapamide) (N=64) | DB Period: Zilebesiran (Add-on to Indapamide) (N=63) | DB Period: Placebo (Add-on to Amlodipine) (N=120) | DB Period: Zilebesiran (Add-on to Amlodipine) (N=118) | DB Period: Placebo (Add-on to Olmesartan) (N=145) | DB Period: Zilebesiran (Add-on to Olmesartan) (N=148) | DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort] (N=26) | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort] (N=63) | DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort] (N=48) | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort] (N=118) | DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort] (N=66) | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort] (N=148) | DB (Placebo) to SFU [Indapamide Cohort] (N=38) | DB (Zilebesiran) to SFU or OLE to SFU [Indapamide Cohort] (N=89) | DB (Placebo) to SFU [Amlodipine Cohort] (N=72) | DB (Zilebesiran) to SFU or OLE to SFU [Amlodipine Cohort] (N=166) | DB (Placebo) to SFU [Olmesartan Cohort] (N=79) | DB (Zilebesiran) to SFU or OLE to SFU [Olmesartan Cohort] (N=214)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in: Indapamide (N=127) | Run-in: Amlodipine (N=238) | Run-in: Olmesartan (N=293) | DB Period: Placebo (Add-on to Indapamide) (N=64) | DB Period: Zilebesiran (Add-on to Indapamide) (N=63) | DB Period: Placebo (Add-on to Amlodipine) (N=120) | DB Period: Zilebesiran (Add-on to Amlodipine) (N=118) | DB Period: Placebo (Add-on to Olmesartan) (N=145) | DB Period: Zilebesiran (Add-on to Olmesartan) (N=148) | DB Period (Placebo) to OLE Period (Zilebesiran) [Indapamide Cohort] (N=26) | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Indapamide Cohort] (N=63) | DB Period (Placebo) to OLE Period (Zilebesiran) [Amlodipine Cohort] (N=48) | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Amlodipine Cohort] (N=118) | DB Period (Placebo) to OLE Period (Zilebesiran) [Olmesartan Cohort] (N=66) | DB Period (Zilebesiran) to OLE Period (Zilebesiran) [Olmesartan Cohort] (N=148) | DB (Placebo) to SFU [Indapamide Cohort] (N=38) | DB (Zilebesiran) to SFU or OLE to SFU [Indapamide Cohort] (N=89) | DB (Placebo) to SFU [Amlodipine Cohort] (N=72) | DB (Zilebesiran) to SFU or OLE to SFU [Amlodipine Cohort] (N=166) | DB (Placebo) to SFU [Olmesartan Cohort] (N=79) | DB (Zilebesiran) to SFU or OLE to SFU [Olmesartan Cohort] (N=214)
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 1 | 4 | 0 | 5 | 0 | 3 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 2 | 6 | 3 | 5 | 1 | 3 | 3 | 9 | 2 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 3 | 8 | 0 | 3 | 1 | 5 | 4 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 3 | 11 | 0 | 3 | 0 | 8 | 3 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 4 | 4 | 5 | 5 | 4 | 0 | 6 | 0 | 6 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 8 | 4 | 16 | 6 | 17 | 14 | 0 | 7 | 3 | 8 | 6 | 14 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05103332/Prot_002.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT05103332/SAP_003.pdf